CLINICAL TRIAL: NCT02302053
Title: A Multi-Center, Randomized, Double-Blind, Placebo-Controlled Clinical Study to Evaluate the Efficacy of the New Viviscal Professional Strength Oral Supplement in Females With Self-Perceived Thinning Hair
Brief Title: Efficacy of the New Viviscal Professional Strength Oral Supplement in Females With Thinning Hair
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ablon Skin Institute Research Center (Other)
Collaborators: Irish Response t/a Lifes2good (Industry); DeNova Research (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: ADHT-0213
Record Dates: First submitted 2014-11-24; First posted 2014-11-26 (Estimated); Last update posted 2014-11-26 (Estimated); Status verified 2014-11

CONDITIONS: Hair Thinning
Keywords: Hair thinning, hair loss, alopecia, women, oral supplement
MeSH Terms: conditions — Alopecia

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- New Viviscal Professional Supplement (Active Comparator): New Viviscal Professional Strength Supplements. One tablet taken by mouth in the morning and one tablet in the evening with food for 180 days.
  Interventions: Dietary Supplement: New Viviscal Professional Supplement
- Placebo Tablet (Placebo Comparator): Placebo tablets. One tablet taken by mouth in the morning and one tablet in the evening with food for 180 days.
  Interventions: Dietary Supplement: Placebo tablets

INTERVENTIONS:
Dietary Supplement: New Viviscal Professional Supplement — The key ingredient is AminoMar C™ marine complex, an organic form of silica derived from Equisetum sp. (horsetail), vitamin C derived from Malpighia emarginata (acerola cherry), microcrystalline cellulose (E460), natural orange flavor, magnesium stearate, hypromellose, and glycerol. The AminoMar C ™ is an active ingredient which has been trademarked and comprises of a proprietary blend of shark powder and mollusc powder. It is derived from sustainable marine sources. Viviscal provides essential nutrients to nourish hair naturally from within. The Viviscal supplement is compared to the placebo tablet which contains no active ingredients. One tablet is taken by mouth in the morning and evening with food.
  Arms: New Viviscal Professional Supplement
Dietary Supplement: Placebo tablets — The placebo tablet contains no active ingredients. One tablet is taken by mouth in the morning and evening with food.
  Arms: Placebo Tablet

SUMMARY:
The New Viviscal Professional Strength is an oral food supplement specifically designed to promote hair growth for women suffering from temporary thinning hair. It does not contain hormones, drugs or industry by-products. Viviscal has been marketed in Europe for over 15 years.

The purpose of this clinical research study is to evaluate certain physiological effects of Viviscal compared to placebo in forty (40) female subjects, ages 21-75 years of age with self-perceived thinning hair associated with poor diet, stress, hormonal influences or abnormal menstrual cycles when compared to using the placebo tablet.

DETAILED DESCRIPTION:
The key ingredient is AminoMar C™ marine complex, an organic form of silica derived from Equisetum sp. (horsetail), vitamin C derived from Malpighia emarginata (acerola cherry), microcrystalline cellulose (E460), natural orange flavor, magnesium stearate, hypromellose, and glycerol. The AminoMar C ™ is an active ingredient which has been trademarked and comprises of a proprietary blend of shark powder and mollusc powder. It is derived from sustainable marine sources. Viviscal provides essential nutrients to nourish hair naturally from within. Viviscal works in 4 stages (see below) over several months of use to improve the appearance of thinning hair.

STAGE 1: Nourishes the hair follicles STAGE 2: Strengthens and promotes the growth of terminal hairs. Terminal hair is defined as coarse hair, short or long, found on the scalp with minimum cross-sectional diameter of 40 micrometers. Vellus hair is defined as fine, short hairs found on the scalp with maximum cross-sectional diameter of 40 micrometers.

STAGE 3: Supports the growth of hair where it has slowed down or temporarily stopped STAGE 4: Hair becomes stronger, healthier and more vibrant

Ingestion of Viviscal over a six (6) month period will strengthen and promote the growth of terminal hairs in female subjects, ages 21-75 years of age with self-perceived thinning hair associated with poor diet, stress, hormonal influences or abnormal menstrual cycles. The primary endpoints will be individual hair counts and favorable analysis using the Nikon CoolPix 4300 with 3GEN Dermlite Foto37 or Nikon D90 camera with a Nikor 105 mm macro lens for phototrichogram analysis at the end of the six (6) month period. The secondary endpoints will be favorable improvements in terminal hair diameter measured by the Dino-Lite Digital Microscopic and positive feedback on the Quality of Life and Self-Assessment questionnaires after six (6) months of Viviscal ingestion.

All patients enrolled must be identifiable throughout the study. The Investigator will maintain a personal list of patient numbers and patient names to enable records to be found at a later date and the list will be stored in a locked cabinet. Subject numbers consist of a 2 digit number from 01 to 40. Patients will be randomized to active or placebo supplements (1:1 ratio) using a randomization table prepared prior to the start of the study by a non-participating staff member at the office of the Investigators. The study blind will not be broken until the end of the study. All test product and placebo will be labeled with subject numbers per the non- participating staff member. Subjects will be assigned a subject number in numerical order as enrolled. Randomization will occur by assignment to either New Viviscal professional strength supplement or placebo with 1:1 ratio. Subjects who terminate their study participation for any reason, regardless of whether study medication was used or not, will retain their randomization number.

Subjects will be assigned a two-digit number which will uniquely identify every subject on the study. This number will remain with the subject throughout the study and should be used in all references to the individual in this study. No number will be reassigned once the study begins. Subjects at the ASIRC will start with 01 to 20 and at DeNova Research 21 to 40. Patients will be identified solely by this number and any paper records which reflect electronic data or relationships of those data with patient confidential information are kept in locked cabinets.

Visit Procedures Pre-Study Procedures

1. Candidate subjects will be screened with the eligibility requirements by telephone prior to Visit 1.
2. Candidate subjects will be assigned an appointment time for visiting the clinic.

Visit 1: Baseline, Day 0

1. Individuals will be given an informed consent (IC) document & photographic release form, HIPAA form, confidentiality agreement to read. They will have all of their study related questions answered by the Investigator or his/her designated staff and if they agree, they will sign two copies of the IC/Photography release form, two copies of the HIPAA form, and one copy of the confidentiality agreement. Subjects will be given one copy of the signed IC/Photography release and of the HIPAA agreement to keep, with one copy of each document remaining at the testing facility in the subject's file.
2. Investigator and/or Study Coordinator will review with subject and complete the checklist for all inclusion and exclusion criteria.
3. Investigator and/or Study Coordinator will review with subject and complete the checklist for medical history and concomitant medications.
4. Investigator and/or Study Coordinator will review with subject and complete the General Lifestyle Questionnaire. The General Lifestyle Questionnaire may be found in Appendix IV.
5. Subjects will be given a Quality of Life Questionnaire to read and complete. The Quality of Life Questionnaire may be found in Appendix V.
6. Candidate subjects will receive a brief physical exam, including examination of the scalp, to rule out any immediately observable medical issues and any scalp alopecias/scalp disorders that are unacceptable for qualification. The physical will additionally include vital signs (pulse and blood pressure), weight and height.
7. Candidate subjects of childbearing potential will complete a urine pregnancy test prior to product distribution.
8. Candidate subjects who have completed all the initial paperwork and meet the inclusion/exclusion qualifications (to include findings of the physical exam) will be assigned a unique subject number. Subjects will be randomized to treatment group prior to dispensing the test product.
9. Qualified subjects will have their scalp prepared for digital photography and initial measurements done (see Appendix I).
10. Subjects will have the selected test site photographed (see Appendix I and II).
11. Subjects will have ten (10) terminal hairs in the selected test site cut at the base of the scalp and the diameter of the hairs measured (see Appendix III).
12. Subjects will be dispensed a three (3) month supply of the test product (three units of Viviscal or Placebo, as randomized, containing 60 tablets each) and given written and verbal Usage and Lifestyle instructions (see Appendix VII) and a calendar of future visits. Subjects will be instructed to ingest the test product per Sponsor instructions.

Usage Instructions:

Take two (2) tablets a day, one in the morning and one in the evening; take with water, after food.

Subjects will be instructed to return all empty packets and unused test product at Visits 2 and 3.

Lifestyle Instructions:

Subjects will be instructed to maintain their normal hair care routine. Subjects will be instructed to use the same brand/type of hair care products and maintain the same haircut, color and style for the study duration.

Subjects who have color treated hair will also be instructed to have the color treatment performed at the same time interval prior to each visit (ie. If on Visit 1, the color treatment was done one week prior then the color treatment is expected to occur at a similar interval of one week prior to Visits 2 and 3).

Subjects will be instructed to come to each visit with clean (shampoo in the morning on the day of the visit) and dry hair.

Subjects will be instructed to use a medically sound form of birth control during the study.

Visit 2: Month 3 (90 days) ± 1 week (7 days)

1. A clinician will ask subjects if they have experienced any changes in their health or taken new/adjusted current medications since the last visit. If an AE or SAE is reported, the examining Investigator will be informed and the appropriate forms will be completed.
2. The test product will be collected and counted for compliance. Subjects found to be consistently out of compliance will be reminded of the correct usage instructions.
3. Subjects will receive a brief physical exam. The physical will include vital signs (pulse and blood pressure).
4. Subjects will complete the Quality of Life Questionnaire and the Self-Assessment Questionnaire (see Appendix V and VI).
5. Subjects will have their scalp prepared for digital photography (see Appendix I).
6. Subjects will have the selected test site photographed (see Appendix I and II).
7. Subjects will have ten (10) terminal hairs in the selected test site cut at the base of the scalp and the diameter of the hairs measured (see Appendix III).
8. Subjects will be dispensed a three (3) month supply of the test product, (three units of Viviscal or Placebo, as randomized, containing 60 tablets each), and given written and verbal Usage and Lifestyle instructions (See Appendix VII). Subjects will be instructed to ingest the test product per Sponsor instructions.

Visit 3: Month 6 (180 days) ± 1 week (7 days)

1. A clinician will ask subjects if they have experienced any changes in their health or taken new/adjusted current medications since the last visit. If an AE or SAE is reported, the examining Investigator will be informed and the appropriate forms will be completed.
2. The test product will be collected and counted.
3. Subjects will receive a brief physical exam. The physical will include vital signs (pulse and blood pressure).
4. Subjects will complete the Quality of Life Questionnaire and the Self-Assessment Questionnaire (see Appendix V and VI).
5. Subjects will have their scalp prepared for digital photography (see Appendix I).
6. Subjects will have the selected test site photographed (see Appendix I and II).
7. Subjects will have ten (10) terminal hairs in the selected test site cut at the base of the scalp and the diameter of the hairs measured (see Appendix III).

All primary and secondary parameters will be collected at Visits 1, 2 and 3. Missing data values will be minimized by intensive training of the interviewers in techniques of clarifying answers and checking questionnaires while participants are on-site. When missing values are identified, several approaches such as rescheduled within 24 hours of completion of tests or interviews will be employed to acquire the necessary data. Missing data will be also examined to assess randomness. Descriptive statistics will be obtained for all variables, tests of normality of continuous measures will be made and data will be examined for homogeneity of variance. An appropriate statistical method will be employed to correct for any abnormalities. All statistical tests will be two-tailed. Differences will be considered statistically significant provided a p-value of 0.05 or less is obtained. For each visit, the differences of the two groups from baseline Visit will be tested using analyses of variance with repeated measurements.

ELIGIBILITY:
Inclusion Criteria:

1. Females, ages 21-75 years of age.
2. Clinically-determined general good health as determined by responses to the initial study assessment.
3. Females with self-perceived thinning hair associated with poor diet, stress, hormone influences or abnormal menstrual cycle as determined on initial study assessment by the Investigator (This will not include patients with medically diagnosed telogen effluvium).
4. Females willing to maintain their normal hair shampooing frequency.
5. Females willing to add the provided oral supplement to their current daily routine.
6. Females willing to not substantially change their current diet, medications, or exercise routines for the duration of the study. If a subject receives physician guidance during the study to change diet, medications, or exercise routine, the subject will need to notify the clinic as soon as possible.
7. Females willing to undergo a brief physical exam to include height, weight, blood pressure, pulse, general physical findings and a scalp exam. The physical exam will occur at Visits 1, 2 and 3.
8. Females with Fitzpatrick I-IV photo skin types.
9. Willingness to have digital photography of the target area and scalp for hair counts at Visits 1, 2 and 3.
10. Willingness to have ten (10) terminal hairs from the target area cut at the base of the scalp for microscopic hair measurements at Visits 1, 2, and 3.
11. Willingness to maintain a consistent hair cut and hair color throughout the 6 month study period and to come to visits with clean (shampoo done in the morning prior to visit) and dry hair.
12. Willingness of subjects who have color treated hair to have the color treatment performed at the same time interval prior to each visit (ie. If on Visit 1 the color treatment was done one week prior then the color treatment is expected to occur at a similar interval of one week prior to Visits 2 and 3)

Exclusion Criteria:

1. Females with a known history of intolerance or allergy to fish, seafood or acerola.
2. Females with any known allergy or sensitivity to any shampoo/conditioner.
3. Females who are nursing, pregnant, planning to become pregnant during the study.
4. Females with known stressful incident within the last six months (ie. death in family, miscarriage)
5. Females who are participating on any clinical research study at ASIRC, DeNova Research or at another research center or doctor's office.
6. Females who have recently (within the last 6 months) started the use of hormones for birth control or hormone replacement therapy (HRT). Women currently using hormones for birth control or HRT must have been on a stable dose (6 months or longer) in order to be eligible for the study.
7. Females currently using the HairMax light treatment or other light therapy to treat thinning hair.
8. Females who have regularly used Rogaine (Minoxidil) within the last 3 months.
9. Females who have used prescription drugs known to affect the hair growth cycle within the last 6 months (e.g., hormone-based birth control for less than 6 months, cyproterone acetate, aldactone/spironolactone, Finasteride or any 5-alpha-reductase inhibitor).
10. Females suffering from other hair loss disorders, such as alopecia areata, scarring alopecia, androgenetic alopecia and telogen effluvium as determined on initial study assessment by the Investigator.
11. Individuals with self-reported uncontrolled diseases (i.e. diabetes, hypertension, hyperthyroidism, hypothyroidism, etc.). Medical conditions that are under control with or without treatment will be considered on an individual basis by the Investigators.
12. Females with self-reported active hepatitis, immune deficiency, HIV or autoimmune disease.
13. Females having a known active dermatologic condition which, in the opinion of the examining Investigators, might place the subject at a greater risk or interfere with clinical evaluations (e.g., seborrheic dermatitis, psoriasis, atopic dermatitis, advanced skin cancer, etc.).

Ages: 21 Years to 75 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2013-02; Primary Completion 2014-02 (Actual); Study Completion 2014-02 (Actual)

PRIMARY OUTCOMES:
Number of terminal hairs in the target area of the scalp. | 180 days
  The first primary efficacy parameter from the phototrichogram will be the number of terminal hairs in the target area of the scalp. Terminal hair is defined as coarse hair, short or long, found on the scalp with minimum cross-sectional diameter of greater than 40 micrometers. Phototrichogram macrophotographs will be taken of the selected target area of each subject at each visit as specified under the Schedule of Procedures. Digital macrophotography will be performed using a Nikon Coolpix 4300 camera with a 3GEN Dermlite Foto37 system for scalp photography. The macrophotographs are then read by the investigator to determine the terminal hair count.
Number of vellus hairs in the target area of the scalp. | 180 days
  The second primary efficacy parameter from the phototrichogram will be the number of vellus hairs in the target area of the scalp. Vellus hair is defined as fine, short hairs found on the scalp with maximum cross-sectional diameter of 40 micrometers. Phototrichogram macrophotographs will be taken of the selected target area of each subject at each visit as specified under the Schedule of Procedures. Digital macrophotography will be performed using a Nikon Coolpix 4300 camera with a 3GEN Dermlite Foto37 system for scalp photography. The macrophotographs are then read by the investigator to determine the vellus hair count.

SECONDARY OUTCOMES:
Dino-Lite microscopic photographs for terminal hair diameter measurements in the target area. | 180 days
  Dino-Lite Microscopic digital photographs to measure the diameter of the hair will be taken of the selected target area of each subject at each visit as specified under the Schedule of Procedures. Ten (10) terminal hairs in the target area will be randomly chosen throughout the area (not all from one direct area) and cut at the surface of the scalp thus not creating any bald patches. The hair diameter will then be measured at 1mm from the cut end of the hair. The ten (10) hair measurements will then be averaged to attain a median hair diameter for the target area.
Quality of Life Questionnaire | 180 days
  Questionnaire about the subjects general lifestyle and how their life is affected by thinning hair.
Self-Assessment Questionnaire | 180 days
  Questionnaire is the evaluation of the growth and qualities related to the subjects hair, nails and skin.

CONTACTS AND LOCATIONS:
Overall Officials: Glynis Ablon, MD, FAAD, Principal Investigator — Director Ablon Skin Institute Research Center; Steven Dayan, MD, FACS, Principal Investigator — Director DeNova Research